CLINICAL TRIAL: NCT06622577
Title: The Effect of Dietary Management and Cysteine Supplementation on Growth Parameters and Biochemical Control for Pediatric Qatari Patients Affected with Classical B6 Non-responsive Homocystinuria.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-23-734
Record Dates: First submitted 2024-07-26; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-07

CONDITIONS: Classical Homocystinuria
Keywords: Methionine; Homocystinuria; cysteine
MeSH Terms: conditions — Homocystinuria | interventions — Cysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dietary management with additional Cysteine supplementation (Experimental)
  Interventions: Dietary Supplement: Cysteine

INTERVENTIONS:
Dietary Supplement: Cysteine — Cysteine supplementation would be given according to the 2001 ROSS guidelines for the HCU. Cys amino acid supplements are available in the form of powder, each sachet containing 4gm which provides 500mg of Cys per sachet that is available in HMC medical store from where patients receive the medical formula and food at free of cost. The dosage of cysteine will be calculated according to the weight of the patient with the age specific recommendation and prescribed by the metabolic dietitian which will be approved by the metabolic physician prior to the supply of cysteine supplements to the patients. It is not known to have any serious adverse events that is life threatening. A single arm interventional study is opted as the intervention involves all the participants without withholding the treatment. Moreover, a single arm interventional study on cysteine supplementation aims to provide evidence on its efficacy contributing to the advancement of clinical practice in HCU management.
  Other Names: single arm interventional study

SUMMARY:
Classical homocystinuria (HCU) is an autosomal recessive disorder caused by the deficiency of an enzyme cystathionine β-synthase (CβS) that affects the catabolic pathway of the amino acid methionine (Met) which leads to an accumulation of high levels of methionine and Homocysteine causing complications in the multi system. Therefore, a strict dietary management is crucial to maintain good biochemical control, growth parameters and avoid complications. The main objective would be to analyze the impact of the Met restricted diet on growth parameters, biochemical markers and long-term complications in patients up to 18 years. In addition, the efficacy of dietary management with additional cysteine (Cys) supplementation for the patients up to 18 years would also be examined.

The participants of the study would be recruited from the metabolic and genetics clinic in Hamad General Hospital (HGH), Qatar. All Qatari participants with confirmed diagnosis of HCU <18 years of age will be included in the study. A mixed method study design would be used which include a cross sectional study design to assess the impact of methionine restricted diet on outcome variables and a single arm interventional study to analyze the effect of additional cysteine supplementation in patients from birth to 18 years. For the retrospective study, all the required data would be retrieved from electronic record from the Cerner of HMC and would be stored in a local drive with password protection. Further, all the eligible participants would be prospectively followed to supplement additional cysteine for the period of 6 months.

The collected data will be statistically analyzed using the "SPSS windows version 22.0 software. The study would improve better understanding of dietary management through the identified outcomes. The outcome of Cys supplementation will improve the protein tolerance, biochemical parameters, growth parameters and may standardize the Cys supplementation.

DETAILED DESCRIPTION:
This single-arm interventional study aims to evaluate the efficacy of dietary management combined with additional cysteine (Cys) supplementation in patients with Classical Homocystinuria (HCU). The study will assess the impact on biochemical markers and growth parameters over a six-month period. The study will include pediatric patients from birth to 18 years old, residing in Qatar, a region with the highest global prevalence of HCU.

Classical HCU is an autosomal recessive disorder resulting from a deficiency in cystathionine β-synthase (CβS). This enzymatic deficiency disrupts the metabolism of methionine (Met) and leads to elevated levels of homocysteine (Hcy), while cysteine (Cys) levels remain low. Untreated, HCU can cause significant complications including ectopic lentis, elongated bones, intellectual disability, and thromboembolism. Management primarily involves dietary restrictions to reduce Met intake and supplementation of Cys, along with other treatments.

More research is needed to determine the appropriate cysteine levels in treated patients and whether additional L-cystine supplementation can improve outcomes in those with Classical homocystinuria.

In CBS deficiency, the formation of cysteine from methionine is disrupted, making cysteine a "conditionally essential" amino acid. Low cysteine concentrations may contribute to the disease's pathogenesis.

The Relationship Between Cysteine and Homocysteine (Hcy) is both cysteine and homocysteine (Hcy) contain thiol groups, and they exist in different reduced and oxidized forms. When Hcy levels are very high, they reduce the concentration of plasma cysteine, likely due to the limited thiol-binding capacity of plasma proteins. Improving homocysteine control by increasing cysteine levels highlights the importance of focusing on cysteine supplementation. Case reports even suggest that cysteine deficiency may lead to poor weight gain and growth, even with adequate energy intake.

Cysteine is added to most methionine-free L-amino acid supplements, but the quantities may not always be sufficient. Administering cysteine can be challenging due to its poor solubility and unpleasant taste.

This provides insight into the complexities of managing CBS deficiency and the potential need for individualized cysteine supplementation.

Despite the known benefits of dietary management, there is limited research on the impact of additional Cysteine supplementation. This study seeks to explore this aspect more comprehensively, especially considering varying practices and guidelines globally.

ELIGIBILITY:
Inclusion Criteria:

* All the patients with a confirmed diagnosis of HCU by molecular and biochemical testing who are either diagnosed through NBS or LD who are following the diet

  * Both male and female gender from birth to 18 years
  * Participants depending on the age of inclusion who are willing to participate

Exclusion Criteria:

* ✔ Patients with Pyridoxine responsive- homocystinuria

  * Patients who are solely on medication without any dietary intervention ✔ Non-Qatari Patients with a confirmed diagnosis of HCU

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
improvement of the biochemical parameters specifically homocysteine and methionine levels | Six months
  Biochemical Parameters:
  Description: The primary outcome will assess the improvement in biochemical parameters, specifically homocysteine (umol/l) and methionine levels(umol/l), in patients with Homocystinuria (HCU) following Cysteine(Cys) supplementation.
  Measurement Tool:
  Blood tests will be used to measure the levels of homocysteine and methionine.

SECONDARY OUTCOMES:
Improvement of growth parameters including weight, Height and BMI | six month
  Growth Parameters:
  Description: The secondary outcome will evaluate changes in growth parameters, including weight, height, and Body Mass Index (BMI), to understand the impact of Cys supplementation on physical growth.
  Weight Measurement:
  Measurement Tool: Standard clinical scales. Unit of Measure: Kilograms (kg)
  Height Measurement:
  Measurement Tool: Stadiometer or measuring tape. Unit of Measure: Centimeters (cm)
  BMI Calculation:
  Calculation: BMI will be calculated using the formula: weight (kg) / height (m²).Unit of Measure: Kilograms per square meter (kg/m²)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of dietetics and Nutrition, Doha, Qatar, Qatar

IPD SHARING:
Plan to Share IPD: No
The country has strict laws preventing sharing of IPD to any third party.